CLINICAL TRIAL: NCT00033748
Title: Sequential Phase II Study of the Anti-Idiotype Monoclonal Antibody Vaccine CeaVac and TriAb in Patients With Minimal Metastatic Colorectal Cancer
Brief Title: Vaccine Therapy in Treating Patients With Colorectal Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-89903; U10CA031946 (NIH); CALGB-89903; CDR0000069324 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Monoclonal Antibody Therapy (Experimental): Patients with minimal metastatic colorectal cancer are treated with 2 anti-idiotype monoclonal antibodies
  Interventions: Biological: monoclonal antibody 11D10 anti-idiotype; Biological: monoclonal antibody 3H1 Alu Gel

INTERVENTIONS:
Biological: monoclonal antibody 11D10 anti-idiotype — 2 mg intradermal injection q 14 days for 4 doses, then sub Q monthly for 4 months, following a 6-12 wk rest period after curative hepatic resection
  Other Names: TriAb
Biological: monoclonal antibody 3H1 Alu Gel — 2 mg intradermal injection q 14 days for 4 doses, then sub Q monthly for 4 months, following a 6-12 wk rest period after curative hepatic resection
  Other Names: CeaVac

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year recurrence-free survival of patients with minimal metastatic colorectal cancer after hepatic resection when treated with adjuvant monoclonal antibody 3H1 anti-idiotype vaccine and monoclonal antibody 11D10 anti-idiotype vaccine.

Secondary

* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Beginning 6-12 weeks after curative hepatic resection, patients receive monoclonal antibody 3H1 anti-idiotype vaccine and monoclonal antibody 11D10 anti-idiotype vaccine intracutaneously at separate sites on days 1, 15, 29, and 45, then subcutaneously monthly for 4 months.

PROJECTED ACCRUAL: A total of 63 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatic colorectal metastases
* Must have undergone complete resection of hepatic colorectal metastases with tumor-free margins (curative resection) at least 6, but no more than 10, weeks prior to study entry
* No evaluable or measurable disease after hepatic resection, documented by intraoperative palpation or imaging studies including intraoperative ultrasound, CT scan, or MRI
* No hereditary non-polyposis colon cancer type B
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 2 mg/dL
* AST no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN

Gastrointestinal:

* No celiac disease
* No familial polyposis
* No Gardner's syndrome
* No Peutz-Jeghers syndrome

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No seizure disorders requiring continuous medication
* No history of clinically significant hypersensitivity reactions, including known hypersensitivity to rodent proteins
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior murine antibodies (e.g., oncoscint scan)
* No prior monoclonal antibody 3H1 anti-idiotype vaccine or monoclonal antibody 11D10 anti-idiotype vaccine

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure or hormones for non-disease-related conditions (e.g., insulin for diabetes)

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* Prior treatment for primary lesion or hepatic metastases allowed
* No concurrent immunomodulatory therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2001-12; Primary Completion 2007-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 2 years

SECONDARY OUTCOMES:
Toxicity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C. Posner, MD, Study Chair — University of Chicago
Locations (75):
- United States (75):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Posner MC, Niedzwiecki D, Venook AP, Hollis DR, Kindler HL, Martin EW, Schilsky RL, Goldberg RM, Mayer RJ. A phase II prospective multi-institutional trial of adjuvant active specific immunotherapy following curative resection of colorectal cancer hepatic metastases: cancer and leukemia group B study 89903. Ann Surg Oncol. 2008 Jan;15(1):158-64. doi: 10.1245/s10434-007-9654-7. Epub 2007 Nov 16. PMID 18008108